CLINICAL TRIAL: NCT06849687
Title: Effect of Whole Body Vibration on Hand Grip Strength, Muscular Activity, and Upper Limb Function in Young Females With Smartphone Addiction: A Randomized Controlled Trial.
Brief Title: Effect of Whole Body Vibration in Young Females With Smartphone Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Assistant Professor of physical therapy for surgery, Faculty of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: No. 7486
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-05

CONDITIONS: Smart Phone Addiction
Keywords: whole body vibration; hand grip strength; muscle activity; upper limb function; smart phone addiction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Whole body vibration group) (Experimental): Whole body vibration (WBV) group will receive vibration on the platform for 20 repetitions in 2 sets with 2 minutes rest between sets in addition to strengthening exercises to the hand muscles.
  Interventions: Device: Whole body vibration; Other: Strengthening exercises
- Group B (Sham Whole body vibration group) (Sham Comparator): participants will receive WBV with the device turned off in addition to strengthening exercises to the hand muscles.
  Interventions: Device: Sham Whole body vibration; Other: Strengthening exercises

INTERVENTIONS:
Device: Whole body vibration — Participants will be asked to sit on an chair without armrests close to the platform and will be asked to perform 90° shoulder flexion, bend both elbows slightly, flex the trunk forwards and place both hands on the platform.
  Arms: Group A (Whole body vibration group)
Device: Sham Whole body vibration — Participants will receive the vibration with the device turned off.
  Arms: Group B (Sham Whole body vibration group)
Other: Strengthening exercises — Participants will use elastic resistance for the finger extension and flexion exercises, and ball to strength wrist flexors for two sets of 10 repetitions within a training session.

SUMMARY:
Young adults have a high prevalence of smartphone addiction. Many adolescents use their smartphones extensively for communication, which starts out as a habit but eventually turns into an addiction. Numerous studies have shown that adolescents use social media for roughly ten hours every day.

ELIGIBILITY:
Inclusion Criteria:

* High smartphone users according to the Smartphone Addiction Scale Short Version (SAS- SV)
* Body mass index (BMI) less than 30 kg/m²
* Didn't receive regular exercise in the last 6 months.

Exclusion Criteria:

* Medical history of median nerve release, hand or thumb tendon lesion
* Prior hand or wrist fractures
* Medical history of hand injuries, and upper limb skin diseases
* WBV contraindications include (joint issues, acute inflammations, back pain, epilepsy, diabetes, or neuromuscular disorders, or dizziness, any discomfort, and nausea)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 4 weeks
  Participants will be asked to perform maximum hand grip with the dominant hand with hold for 5 seconds, for three repetitions using the hand held dynamometer (dynamometer, Jamar, United States), a 60 seconds rest interval will be planned in between the repetitions. The mean of the three repetitions will used for calculation of hand grip strength.

SECONDARY OUTCOMES:
pinch strength | 4 weeks
  The participant will be asked to sit comfortably, with the pinch gauge between the index and middle fingers, and thumb, with the tested arm at the side with the elbow flexed 90 degrees. After five seconds of holding the pinch with full force, take a reading, repeat three times.
Muscle activity of flexor carpi radialis muscle | 4 weeks
  Muscle activity will be measured utilizing electromyography (EMG) using the Delsys Trigno (DST01) system for flexor carpi radialis muscle.
Muscle activity for flexor carpi ulnaris muscle | 4 weeks
  Muscle activity will be measured utilizing electromyography (EMG) using the Delsys Trigno (DST01) system for flexor carpi ulnaris muscle.
Muscle activity for extensor digitorum communis muscle | 4 weeks
  Muscle activity will be measured utilizing electromyography (EMG) using the Delsys Trigno (DST01) system for extensor digitorum communis muscle.
Upper limb function | 4 weeks
  The upper limb function will be assessed by using the Arms, Shoulders and Hands Disability Questionnaire (DASH) Quick, which is a validated and widely used 11-item questionnaire that evaluates certain impairments and symptoms in the upper limb. the score ranged from 0 to 100, the lower the score, the greater the results. While, higher scores represent the worst results.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol